CLINICAL TRIAL: NCT01370109
Title: The Cardiovascular Effects of Sunitinib Therapy: Off Target Changes in Cardiac Metabolism and Ventricular Vascular Mechanics (CREST)
Brief Title: Cardiovascular Effects of Sunitinib Therapy (CREST)
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 34810
Record Dates: First submitted 2011-05-26; First posted 2011-06-09 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Renal Cell Carcinoma 4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Penn Site: Patients with renal cell cancer newly undergoing therapy with the oral tyrosine kinase inhibitor sunitinib will be recrutied and observed over a period of approximately 33 weeks, with additional follow-up at 1 and 2 years.
- Vanderbilt University Medical Center: Patients with renal cell cancer newly undergoing therapy with the oral tyrosine kinase inhibitor sunitinib will be recrutied and observed over a period of approximately 33 weeks.
- Case Medical Center: Patients with renal cell cancer newly undergoing therapy with the oral tyrosine kinase inhibitor sunitinib will be recrutied and observed over a period of approximately 33 weeks.
- University of Wisconsin at Madison: Patients with renal cell cancer newly undergoing therapy with the oral tyrosine kinase inhibitor sunitinib will be recrutied and observed over a period of approximately 33 weeks.

SUMMARY:
Tyrosine kinase inhibitors such as sunitinib are used in the treatment of renal cell carcinoma and have significant off-target effects with cardiac toxicity and resultant ventricular cardiac dysfunction being a major concern. However, the mechanisms of these effects in humans remains poorly defined, as are the clinical methods to risk stratify and identify patients who will ultimately suffer from cardiac dysfunction. The goal of this multi-center study is to characterize the cardiovascular measures of cardiac function; 2) comprehensive measures of arterial function and left ventricular afterload; 3) biomarkers reflective of the pathophysiologic alterations. Through this work, the investigators will translate our basic understanding of sunitinib cardiotoxicity to humans and identify early predictors of sunitinib cardiotoxicity.

DETAILED DESCRIPTION:
Tyrosine kinase inhibitors such as sunitinib have dramatically improved the overall management of certaincancers including renal cell carcinoma. However, recent data suggest that these therapieshave significant off-target effects with cardiac toxicity, including significant hypertension and ventricular cardiac dysfunction being a major concern. However, the biologic mechanisms underlying cardiotoxicty in humans remain poorly defined. Moreover, there is a critical need to develop methods to improve the risk stratification and early identification of patients who will suffer from hypertension and cardiac dysfunction with exposure to therapy. The over all objectives ofthis study are to further characterize the cardiovascular changes that occur with sunitinib exposure in order to improve our understanding of sunitib toxicity and determine early, mechanistically and clinically relevant predictors to identify patients at increased risk of hyptertension and cardiac dysfunction. The specific aims of this study are: 1) To define the changes in arterial hemodynamics that may occur with exposure to sunitinib, 2) To define the changes in sensitive echocardiographic measures of cardiac function that may occur with exposure to sunitinib, 3) To determine blood markers that are associated with changes in vasculature or cardiac function with exposure to sunitinib. and 4) To determine if there are early imaging or biomarker predictors of subitinib cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal cell carcinoma newly undergoing therapy with sunitinib.
* Age greater than or equal to 18 years
* ECOG performance status 0,1,2

Exclusion Criteria:

* Any contraindication to sunitinib therapy of note, patients with prior cardiovascular history are not excluded from this study, as long as there are no contraindications to sunitinib therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our target population is patients with renal cell carcinoma who are newly initiating therapy with the oral tyrosine-kinase inhibitor sunitinib.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure | 6 Months

SECONDARY OUTCOMES:
Number of Participants with adverse events | 2 years
  Number of subjects with adverse events specifically, incident of hypertension and Cardiac dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, Principal Investigator — Abramson Cancer Center at the University of Pennsylvania
Locations (1):
- Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania, United States